CLINICAL TRIAL: NCT06501248
Title: Effect of Triticum Aestivum vs Placebo on Metabolic Profile Components and Insulin Sensitivity in Patients With Obesity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2022-1301-178
Record Dates: First submitted 2024-03-26; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2023-08

CONDITIONS: Obesity; Drug Effect; Insulin Sensitivity
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial, of two parallel groups, double blind, with random assignment and control group.
  36 patients:
  1. 18 patients with 500 mg of triticum aestivum orally every 12 hours for 120 days.
  2. 18 patients with 500 mg of placebo orally every 12 hours for 120 days.
     * Visit 1/ Day -7: Screening period, information about the study, signing of informed consent, medical history, anthropometric measurements, baseline laboratory tests.
     * Visit 2/Day 0: Randomization, 60 tablets of Triticum aestivum or placebo will be given, general diet and exercise recommendations.
     * Visit 3,4,5/Day 30,60,90: Treatment adherence evaluation, laboratory tests, adverse events evaluation, general diet and exercise recommendations and 60 tablets of Triticum aestivum or placebo will be given.
     * Visit 6 /Final/Day 120 ± 7: Anthropometric measurements will be taken, laboratory tests will be performed, adherence to treatment and adverse events will be evaluated.
Who Masked: Participant, Investigator
Masking Description: All participants will be submitted to the selection of a sealed envelope which will have a numerical code previously defined by a third party for each intervention group.
  The total number of envelopes required to complete the minimum number of participants will have numerical codes that identify the bottle of intervention treatment that should receive the participant during the intervention period.
  They will be divided into half blinded codes for triticum aestivum group and half for placebo to complete the size of each subsample. Chance guarantees blinding, neither the participant nor the researcher will know the type of treatment. The database for the blinded statistical analysis will be completed. The blind man will be removed once the statistical analysis has been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triticum aestivum (Active Comparator): A group of 18 patients with a diagnosis of obesity without pharmacological or surgical treatment, who will receive 500 mg of triticum aestivum orally every 12 hours for 120 days.
  Interventions: Drug: Triticum Aestivum
- Placebo (calcined magnesia) (Placebo Comparator): A group of 18 patients diagnosed with obesity without pharmacological or surgical treatment, who will receive 500 mg of placebo (calcined magnesia) orally every 12 hours for 120 days.
  Interventions: Drug: Placebo (calcined magnesia)

INTERVENTIONS:
Drug: Triticum Aestivum — The intervention period will be 120 days, searching for effects on insulin sensitivity and metabolic control.
  Arms: Triticum aestivum
Drug: Placebo (calcined magnesia) — The intervention period will be 120 days, searching for effects on insulin sensitivity and metabolic control.
  Other Names: Calcined magnesia
  Arms: Placebo (calcined magnesia)

SUMMARY:
Obesity is a metabolic disease which has been declared as the most prevalent chronic health problem in adults; according to the World Health Organization (WHO), it is defined as an increase in Body Mass Index (BMI) greater than or equal to 30 kg/m2.

In Mexico, according to data from the National Health and Nutrition Survey (ENSANUT) 2018-2019, the prevalence of overweight in adults is 39.1% (36.6% in women, 42.5% in men), of obesity is 36.1% (40.2% in women, 30.5% in men) and of abdominal adiposity 81.6% (88.4% in women and 72.1% in men), with a higher proportion found in the north of the country.

In 2010, it was estimated that obesity was the main cause of 3.4 million deaths, the main complications being cardiovascular disease, diabetes mellitus and various types of cancer.

The complications of obesity are very varied, mainly presenting changes in the metabolic profile, such as increased blood pressure and abdominal circumference, hypertriglyceridemia and hypercholesterolemia. Another of the main complications derived from obesity is insulin resistance, which is defined as a decreased biological response of peripheral tissues to a specific concentration of insulin with consequent compensatory hyperinsulinemia.

The treatment of obesity is based on lifestyle changes (diet and exercise), in addition, there are pharmacological and surgical treatments, however, they are not applicable to the entire population, so despite being a highly prevalent disease with major complications, current therapeutic options are insufficient.

Triticum aestivum, better known as wheat grass, is a very common fiber in the diet of the world population, including the Mexican population, in which multiple pre-clinical studies have been reported where the effect of triticum aestivum on the decrease of components of the metabolic profile, such as glycemia, cholesterol, triglycerides and weight, as well as an improvement in insulin sensitivity, has been evidenced; To date, no serious adverse effects related to its consumption have been described, and it can be considered as an effective therapeutic alternative for patients with obesity.

DETAILED DESCRIPTION:
A double-blind clinical trial is proposed, with two parallel groups, with random assignment and group control. The universe of the sample will be patients with a diagnosis of obesity, residents of the Guadalajara Metropolitan Area, who agree to participate by signing informed consent and can go to the Biomedical Unit 02 of the Mexican Institute of Social Security. A total of 36 patients will be followed, which will be distributed as follows: 1) A group of 18 patients with a diagnosis of obesity without pharmacological or emergency treatment, who will receive 500 mg of triticum aestivum orally every 12 hours for 120 days, and 2) A group of 18 patients diagnosed with obesity without pharmacological or surgical treatment, who will receive 500 mg of placebo (calcined magnesia) orally every 12 days for 120 days.

ELIGIBILITY:
Inclusion Criteria:

* Ability to communicate and meet all study requirements.
* People who sign the consent under written information prior to carrying out any procedure
* People of any sex, (eumenorrheic women with mechanical or definitive contraceptive method without hormonal treatment) Mexicans from 30 to 50 years of age, residents of Guadalajara, Jalisco, beneficiaries of the Instituto Mexicano del Seguro Social (IMSS)
* People with a diagnosis of Obesity (BMI ≥30 - 39.9 kg/m2), stable body weight within the 3 months prior to the start of the study, defined as a variability in body weight of less than 5%.
* Fasting glucose <126 mg/dl
* Cholesterol <240 mg/dl
* Triglycerides <300 mg/dl
* Resting systolic blood pressure less than 140 mmHg with resting diastolic blood pressure less than 90 mmHg

Exclusion Criteria:

* Suspected or confirmed pregnancy.
* Women breastfeeding or in the postpartum or postpartum period.
* History of smoking at any intensity within the 12 months prior to the start of the study.
* Excessive sedentary lifestyle defined as physical activity less than the equivalent of 15 minutes of walking per day.
* Excessive exercise, defined as physical activity equivalent to running for 60 minutes a day.
* Intake of drugs that are anorexigenic, lipid-lowering or have an effect on body weight.
* History of any type of cancer, hyperthyroidism, hypothyroidism, kidney disease, liver disease, and pancreatic disease.
* History of hypersensitivity to the study drug (gluten)
* History of drug intake
* Carrying of a pacemaker, or any other permanent bioelectronic element that can modify the electrical bioimpedance reading or can be affected by it.
* Patients diagnosed with Morbid Obesity (BMI ≥ 40 kg/m2)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
The effect of Triticum aestivum on glucose in patients with obesity | 120 days
  Changes in levels of glucose in mg/dl.
The effect of Triticum aestivum on insulin sensitivity in patients with obesity | 120 days
  Changes in levels of insulin sensitivity in the triglyceride and glucose index (natural logarithm ((glucose in mg/dl * triglycerides in mg/dl)/2))
The effect of Triticum aestivum on high-density lipoprotein cholesterol in patients with obesity | 120 days
  Changes in levels of high-density lipoprotein in mg/dl.
The effect of Triticum aestivum on low-density lipoprotein cholesterol in patients with obesity | 120 days
  Changes in levels of low-density lipoprotein cholesterol in mg/dl.
The effect of Triticum aestivum on very low-density lipoprotein cholesterol in patients with obesity | 120 days
  Changes in levels of very low-density lipoprotein cholesterol in mg/dl.
The effect of Triticum aestivum on total cholesterol in patients with obesity | 120 days
  Changes in levels of total cholesterol in mg/dl.
The effect of Triticum aestivum on triglycerides in patients with obesity | 120 days
  Changes in levels of triglycerides in mg/dl.
The effect of Triticum aestivum on body weight in patients with obesity | 120 days
  Changes in levels of body weight in kilograms.
The effect of Triticum aestivum on Body Mass Index in patients with obesity | 120 days
  Changes in levels of Body Mass Index (weight in kilograms / (height in meters squared))
The effect of Triticum aestivum on fat percentage in patients with obesity | 120 days
  Changes in levels of fat percentage (percentage)
The effect of Triticum aestivum on Waist Hip Index in patients with obesity | 120 days
  Changes in levels of Waist Hip Index (waist in centimeters / hip in centimeters)

SECONDARY OUTCOMES:
The effect of Triticum aestivum on blood pressure in patients with obesity | 120 days
  Changes in levels of blood pressure in mmHg.
The effect of Triticum aestivum on renal profile in patients with obesity | 120 days
  Changes in levels of creatinine in mg/dl.
The effect of Triticum aestivum on hepatic profile in patients with obesity | 120 days
  Changes in levels of Alanine aminotransferase in mg/dl and Aspartate aminotransferase in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Sandra O Hernández González, PhD, Principal Investigator — Instituto Mexicano del Seguro Social, Unidad de Investigación Biomédica 02
Locations (1):
- Biomedical Unit Research 02, Specialties Hospital, Medical Unit of High Specialty, West National Medical Center, Mexican Social Security Institute., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All data resulting from the clinical investigation, except the personal identification of the subjects (name, address, telephone, etc.)
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication.
Access Criteria: The data can be shared through a request addressed to the principal investigator Dr. Sandra Ofelia Hernández González, basing the reason for what they are requested.

REFERENCES:
- [Background] Kim SY. The Definition of Obesity. Korean J Fam Med. 2016 Nov;37(6):309. doi: 10.4082/kjfm.2016.37.6.309. Epub 2016 Nov 18. No abstract available. PMID 27900066
- [Background] Aktar N, Qureshi NK, Ferdous HS. Obesity: A Review of Pathogenesis and Management Strategies in Adult. Delta Medical College Journal. 2017 Feb 4; 5(1):35-48.
- [Background] Barquera S, Hernandez-Barrera L, Trejo-Valdivia B, Shamah T, Campos-Nonato I, Rivera-Dommarco J. [Obesity in Mexico, prevalence andtrends in adults. Ensanut 2018-19.]. Salud Publica Mex. 2020 Nov-Dec;62(6):682-692. doi: 10.21149/11630. Spanish. PMID 33620965
- [Background] Moreno-Altamirano L, García-García JJ, Soto-Estrada G, Capraro S, Limón-Cruz D. Epidemiología y determinantes sociales asociados a la obesidad y la diabetes tipo 2 en México. Revista Médica Del Hospital General De México. 2014 Jul; 77(3):114-23.
- [Background] Bihan H, Choleau C, Cohen R, Reach G. [Obesity, immune resistance and metabolic complications: what morbid obesity can teach the doctor]. Presse Med. 2007 Dec;36(12 Pt 3):1893-7. doi: 10.1016/j.lpm.2007.04.001. Epub 2007 Apr 24. French. PMID 17459653
- [Background] Ahmed B, Sultana R, Greene MW. Adipose tissue and insulin resistance in obese. Biomed Pharmacother. 2021 May;137:111315. doi: 10.1016/j.biopha.2021.111315. Epub 2021 Feb 6. PMID 33561645
- [Background] Roberts CK, Hevener AL, Barnard RJ. Metabolic syndrome and insulin resistance: underlying causes and modification by exercise training. Compr Physiol. 2013 Jan;3(1):1-58. doi: 10.1002/cphy.c110062. PMID 23720280
- [Background] D'Adamo E, Caprio S. Type 2 diabetes in youth: epidemiology and pathophysiology. Diabetes Care. 2011 May;34 Suppl 2(Suppl 2):S161-5. doi: 10.2337/dc11-s212. No abstract available. PMID 21525449
- [Background] Almeda-Valdes P, Bello-Chavolla OY, Caballeros-Barragan CR, Gomez-Velasco DV, Viveros-Ruiz T, Vargas-Vazquez A, Aguilar-Salinas CA. [Indices para la evaluacion de la resistencia a la insulina en individuos mexicanos sin diabetes]. Gac Med Mex. 2018;154(Supp 2):S50-S55. doi: 10.24875/GMM.18004578. Spanish. PMID 30532124
- [Background] Guerrero-Romero F, Simental-Mendia LE, Gonzalez-Ortiz M, Martinez-Abundis E, Ramos-Zavala MG, Hernandez-Gonzalez SO, Jacques-Camarena O, Rodriguez-Moran M. The product of triglycerides and glucose, a simple measure of insulin sensitivity. Comparison with the euglycemic-hyperinsulinemic clamp. J Clin Endocrinol Metab. 2010 Jul;95(7):3347-51. doi: 10.1210/jc.2010-0288. Epub 2010 May 19. PMID 20484475
- [Background] Rodrigo-Cano S, Soriano Del Castillo JM, Merino-Torres JF. Causas y tratamiento de la obesidad. Nutricion Clinica y Dietetica Hospitalaria. 2017; 37(4):87-92.
- [Background] Fonseca-Junior SJ, Sa CG, Rodrigues PA, Oliveira AJ, Fernandes-Filho J. Physical exercise and morbid obesity: a systematic review. Arq Bras Cir Dig. 2013;26 Suppl 1:67-73. doi: 10.1590/s0102-67202013000600015. English, Portuguese. PMID 24463903
- [Background] Daneschvar HL, Aronson MD, Smetana GW. FDA-Approved Anti-Obesity Drugs in the United States. Am J Med. 2016 Aug;129(8):879.e1-6. doi: 10.1016/j.amjmed.2016.02.009. Epub 2016 Mar 4. PMID 26949003
- [Background] Kushner RF. Weight Loss Strategies for Treatment of Obesity: Lifestyle Management and Pharmacotherapy. Prog Cardiovasc Dis. 2018 Jul-Aug;61(2):246-252. doi: 10.1016/j.pcad.2018.06.001. Epub 2018 Jun 8. PMID 29890171
- [Background] Moshawih S, Abdullah Juperi RNA, Paneerselvam GS, Ming LC, Liew KB, Goh BH, Al-Worafi YM, Choo CY, Thuraisingam S, Goh HP, Kifli N. General Health Benefits and Pharmacological Activities of Triticum aestivum L. Molecules. 2022 Mar 17;27(6):1948. doi: 10.3390/molecules27061948. PMID 35335312
- [Background] Singh N, Verma P, Pandey BR. Therapeutic Potential of Organic Triticum aestivum Linn. (Wheat Grass) in Prevention and Treatment of Chronic Diseases: An Overview [Internet]. Vol. 4, International Journal of Pharmaceutical Sciences and Drug Research. 2012. Available from: www.ijpsdr.com
- [Background] Anup S. PHYTOCHEMICAL AND PHARMACOLOGICAL SCREENING OF WHEATGRASS JUICE (TRITICUM AESTIVUM L.). International Journal of Pharmaceutical Sciences Review and Research. 2011; 9(1):159-64.
- [Background] Leoncini E, Prata C, Malaguti M, Marotti I, Segura-Carretero A, Catizone P, Dinelli G, Hrelia S. Phytochemical profile and nutraceutical value of old and modern common wheat cultivars. PLoS One. 2012;7(9):e45997. doi: 10.1371/journal.pone.0045997. Epub 2012 Sep 26. PMID 23049918
- [Background] Luyen BT, Thao NP, Tai BH, Lim JY, Ki HH, Kim DK, Lee YM, Kim YH. Chemical constituents of Triticum aestivum and their effects on adipogenic differentiation of 3T3-L1 preadipocytes. Arch Pharm Res. 2015 Jun;38(6):1011-8. doi: 10.1007/s12272-014-0478-2. Epub 2014 Sep 23. PMID 25241774
- [Background] Amira Moheb T. Biochemical, Molecular and Pharmacological Studies of the Wheat (Triticum aestivum L). 2012.
- [Background] Kothari S, Jain AK, Mehta SC, Tonpay SD. Hypolipidemic effect of fresh Triticum aestivum (wheat) grass juice in hypercholesterolemic rats. Acta Pol Pharm. 2011 Mar-Apr;68(2):291-4. PMID 21485304
- [Background] Mohan Y, Jesuthankaraj GN, Ramasamy Thangavelu N. Antidiabetic and Antioxidant Properties of Triticum aestivum in Streptozotocin-Induced Diabetic Rats. Adv Pharmacol Sci. 2013;2013:716073. doi: 10.1155/2013/716073. Epub 2013 Dec 14. PMID 24416041
- [Background] Shakya G, Randhi PK, Pajaniradje S, Mohankumar K, Rajagopalan R. Hypoglycaemic role of wheatgrass and its effect on carbohydrate metabolic enzymes in type II diabetic rats. Toxicol Ind Health. 2016 Jun;32(6):1026-32. doi: 10.1177/0748233714545202. Epub 2014 Aug 12. PMID 25116122
- [Background] Im JY, Ki HH, Xin M, Kwon SU, Kim YH, Kim DK, Hong SP, Jin JS, Lee YM. Anti-obesity effect of Triticum aestivum sprout extract in high-fat-diet-induced obese mice. Biosci Biotechnol Biochem. 2015;79(7):1133-40. doi: 10.1080/09168451.2015.1006567. Epub 2015 Apr 30. PMID 25925980
- [Background] Ajiboye BO, Oloyede HOB, Salawu MO. Antidiabetic Activity of Triticum aestivum Seed-Based Diet on Alloxan-Induced Diabetic Rats. J Diet Suppl. 2020;17(2):133-149. doi: 10.1080/19390211.2018.1492485. Epub 2018 Oct 4. PMID 30285545